CLINICAL TRIAL: NCT04443361
Title: Insomnia After the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Sverre Urnes Johnson, Associate Professer Sverre Urnes Johnson, University of Oslo
Other Study IDs: REK125510 (7)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Insomnia; Metacognitive Beliefs; Anxiety; Depression; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the levels of insomnia 3 months after (T2) the strict physical distancing government initiated physical distancing protocols related to the COVID-19 pandemic (T1). The study also aims to investigate how predictors measured after and before the COVID-19 pandemic are associated with sleep problems at T2.

DETAILED DESCRIPTION:
Hypothesis/Research Questions H1: What is the level of mental insomnia following three months of strict mitigation strategies (i.e., physical distancing) in the general adult population during the COVID-19 pandemic? The mean level of insomnia will be benchmarked against the mean level of insomnia in similar pre-pandemic samples.

Exploratory: What is the level of insomnia in different demographic subgroups.

H2: The level of metacognition, strategies, worry about job and economy, health-anxiety and physical activity at T2 will predict insomnia at T2, beyond and above, age, gender, and education.

Exploratory: Does metacognition, strategies, worry about job and economy, health-anxiety and physical activity at T1 predict Insomnia at T2, beyond and above psychiatric diagnosis, age, gender, and education and predictors at T2?

Statistical analysis:

A hierarchical regression analysis will be conducted using BIS as the dependent variable. In the first step stable characteristics (control variables) will be included: age, gender and education. In the second step metacognition, strategies, worry about job and economy, health-anxiety and physical activity at T2 will be included. Part-correlation will be reported for step 2, presenting the effect size of the predictors on insomnia. In the third step, anxiety and depression at T2 will be included as control for the variables at the next step. In the last step metacognition, strategies, worry about job and economy, health-anxiety and physical activity, at T1 will be included.

Multicollinearity and other statistical assumptions will be checked. Multicollinearity will be assessed with common guidelines (VIF < 5 and Tolerance > 0.2; Hocking, 2003; O'Brian, 2007). Descriptive statistics with frequency tables including N, means and SDs and other standard descriptive statistics will be used to examine the level of insomnia. Subgroup differences will be examined with chi-squared statistics or other statistic based on the characteristics of the data (e.g. skewness).

All analysis and questions addressed in the forthcoming paper that are not pre-specificd in this pre-registered protocol will be defined as exploratory.

Sensitivity analyses and random subsample replications of the main finding will be conducted following selection of a random sample of participants that ensure a proportional ratio between the collected sample and the adult population in Norway

Measures On the CAS1 four items were combined into the subscale "positive metacognition", four items were combined into the subscale "negative metacognition", and 8 items were combined into the subscale strategies (Nordahl & Wells, 2019). Physical activity was measured with a single item. Worry about job and economy consisted of two items. Health anxiety consists of four items.

Possible transformations:

All variables will be assessed in their original and validated format as is recommended practice, as long as this is possible with regards to statistical assumptions underlying the pre-defined analyses (i.e., multiple regression). However, if this is not possible with regards to the statistical assumptions behind the analyses, transformation (e.g., square root or log-transformations) may be needed to apply interval-based methods, alternatively the use of non-parametric tests.

Inference criteria Given the large sample size in this study, the investigators pre-define their significance level: p < 0.01 to determine significance.

Sample size:

The present study is part of a larger project with the part aiming to investigate predictors of sleep trough regression analysis, and the second part aiming to examine directional relations among specific symptoms and their centrality through network analysis. Thus, the power calculations are based on power required for network analysis.

Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants are three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. Thus, following these two approaches respectively, between 1584 to 5280 participants are required. Data will be collected for three weeks, and participants are based on a representative and random sample of Norwegian adults, randomly selected and provided equal opportunity to partake in the study, providing digital consent.

Eligibility criteria:

Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who had provided digital consent to partake in the study.

Exclusion Criteria:

• Children and adolescents (individuals below 18) Adults not residing in Norway during the measurement period

Missing data:

The TSD system (Services for Sensitive Data), a platform used in Norway to store person-sensitive data verifies participants officially through a kind of national ID number to give them full right to withdraw their data at any time, following the European GDPR (General Data Protection Regulation) laws. Accordingly, participants are allowed to withdraw their own data at any time. The survey includes mandatory fields of response. Participation is voluntarily, and withdrawal of provided data is possible at any moment. We do not expect participants to withdraw their data and thus expect no missing data. However, if participants do withdraw their data, we will conduct state-of-art missing data analyses and investigate whether data is missing at random.

Exploratory:

Questions addressed in the future paper which is not pre-specified will be defined as exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who had provided digital consent to partake in the study.

Exclusion Criteria:

• Children and adolescents (individuals below 18) Adults not residing in Norway during the measurement period

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The general population in Norway.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
Bergen insomnia scale (BIS) | Data is set to be collected starting from 22th of June. The data collection period will last no longer than three weeks depending on the response to the questionnaire
  Bergen Insomnia scale is developed as a short measure of insomnia consisting of six items measured on a 8-point Likert-scale (Pallesen et al., 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Asle Hoffart, PhD, Principal Investigator — University of Oslo & Modum Bad; Omid Ebrahimi, Mr, Principal Investigator — University of Oslo & Modum Bad; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo & Modum Bad

IPD SHARING:
Plan to Share IPD: No